CLINICAL TRIAL: NCT03403686
Title: LXR as a Novel Therapeutic Target in DR
Brief Title: Liver X Receptor (LXR) as a Novel Therapeutic Target in Diabetic Retinopathy (DR)
Acronym: LXR and DR
Status: Recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria Grant, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: 300000068
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Retinopathy
Keywords: Liver X receptor; Circulating angiogenic cells
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Controls: Any man or woman between the ages of 21- 98 years of age will be eligible to participate. To participate in the study as a study subject we will require that the subject must carry the diagnosis of healthy control.
  Interventions: Biological: blood draw
- Diabetic no retinopathy: Patients with diabetes but with no evidence of diabetic retinopathy
  Interventions: Biological: blood draw
- Diabetic with mild retinopathy: Diabetics with mild non proliferative diabetic retinopathy (NPDR).
  Interventions: Biological: blood draw
- Diabetic with moderate retinopathy: Diabetics with moderate NPDR
  Interventions: Biological: blood draw
- Diabetics with severe retinopathy: Diabetic with severe NPDR.
  Interventions: Biological: blood draw
- Diabetics with proliferative diabetic retinopathy (PDR): Diabetics with proliferative diabetic retinopathy (PDR)
  Interventions: Biological: blood draw

INTERVENTIONS:
Biological: blood draw — Blood sample will be obtained and CD34+ cells will be isolated for functional testing.

SUMMARY:
Results from large clinical trials demonstrate a strong association between lipid abnormalities and progression of the most common microvascular complication, diabetic retinopathy (DR). We found that activation of a master regulator of cholesterol metabolism, the nuclear hormone receptors liver X receptors (LXRα/LXRβ), prevents DR in rodent models. In this application, we seek to understand the mechanisms responsible for the beneficial effects of LXR agonists on retina and on bone marrow (BM) to preserve the function of reparative cells while reducing inflammatory cell.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is a disabling microvascular complication. Despite recent advances using pharmacotherapy, a cure for DR has yet to be realized. Thus, a conceptual and technical breakthrough to identify novel targets, and a strategy to cure this complication is paramount. We believe that the recent clinical evidence from large clinical trials demonstrating a strong association between lipid abnormalities and DR progression and the discovery that activation of the nuclear hormone receptors liver X receptors (LXRα/LXRβ) prevents DR in rodent models offers such a breakthrough. The detrimental effect of dyslipidemia is not limited to the vasculature but also leads to dysfunction of circulating angiogenic cells (CAC) and of macrophages. The endogenous ligands for LXRs are oxidative metabolites of cholesterol that serve as intracellular cholesterol "sensors". LXR agonists operate, in part, by transcriptional upregulation of genes involved in promoting cholesterol efflux and inhibition of cholesterol uptake; and by inhibiting inflammation. Our published studies and new preliminary data show that pharmacological LXR activation prevents DR development in both T1D and T2D rodent models. In this application, we seek to understand the mechanisms involved in this beneficial effect. We put forth the hypothesis that LXR activation will restore cholesterol homeostasis in the diabetic retina and correct diabetes-induced bone marrow dysfunction to sustain CAC levels and function and to reduce of myeloid cell production.

ELIGIBILITY:
Inclusion Criteria:

* Any man or woman between the ages of 21- 98 years of age will be eligible to participate. To participate in the study as a study subject we will require: a) the subject must either carry the diagnosis of diabetes or be a healthy aged control and b) the patient be willing and have the ability to cooperate with the protocol.

Exclusion Criteria:

* Exclusion criteria: We will apply the following exclusion criteria: a) evidence of ongoing acute or chronic infection (HIV, Hepatitis B or C, tuberculosis); b) ongoing malignancy; c) cerebral vascular accident or cerebral vascular procedure; d) current pregnancy; e) history of organ transplantation; f) presence of a graft (to avoid any effect of the graft on inflammatory parameters; g) uremic symptoms, an estimated glomerular filtration rate of less than 20 cc/min (by Modification of Diet in Renal Disease equation), or an albumin of less than 3.6 (to avoid malnutrition as a confounding variable); h) be unwilling to abstain from drinking alcohol and i) patients with anemia. Subjects with AMD, glaucoma, uveitis, known hereditary degenerations or other significant ocular complications other than diabetic retinopathy will be excluded.

Ages: 21 Years to 98 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have retinal abnormalities other than diabetic retinopathy will be excluded. Patients who have systemic conditions that influence hematopoietic stem cell function such as cardiovascular disease, malignant disease, diabetes, hematologic disorder, or estimated glomerular filtration rate less than 60 mL/min or who have undergone treatment with erythropoietin will be excluded. We will record all medications including antihypertensive drug treatment, treatment with statins, Angiotensin-Converting Enzyme (ACE) Inhibitors, Angiotensin Receptor Blockers (ARB) or other pharmacological agents that may influence CD34+ cell function. Baseline characteristics will be recorded, including age, lipid parameters, body mass index (BMI), blood pressure, smoking history, antioxidant intake and use of nutritional supplements.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessing CD34+ cells function | from blood draw to 48 hours
  We are isolating CD34+ cells from peripheral blood and then examining the cell membrane characteristics of CD34+ cells and their in vitro function.

CONTACTS AND LOCATIONS:
Overall Officials: Maria B Grant, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No